CLINICAL TRIAL: NCT05930899
Title: Translational-Omics in Aortic Stenosis (TOmAS) Biobank
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, George Thanassoulis, Professor of Medicine, Director, Preventive and Genomic Cardiology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: A02-M104-13A
Record Dates: First submitted 2023-06-22; First posted 2023-07-05 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases; Aortic Valve Stenosis
MeSH Terms: conditions — Cardiovascular Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biological material including plasma, saliva, genetic material (DNA, RNA, etc.), and tissue explanted during surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CVD Group: CVD diagnosis including, but not limited to: Aortic Stenosis, Coronary Heart Disease, Heart Failure, Atrial Fibrilation, Dilated Cardiomyopathy, Myocardial Infarction, and Spontaneous Coronary Artery Dissection.
  Interventions: Other: Genetics
- Control Group: control groups will be defined as:
  1. No echocardiographic evidence of AS (or any aortic valve abnormality) and
  2. 60 years of age
  Interventions: Other: Genetics

INTERVENTIONS:
Other: Genetics — TOmAS is a biobank and all patients will be genotyped

SUMMARY:
The objective of the TOmAS Biobank is the conservation of biological material (plasma, saliva, and tissue explanted during surgery), genetic material (DNA, RNA, etc.), and clinical data ("material/data") collected from patients with cardiovascular diseases (CVD) as well as from control participants, in order to allow future studies evaluating novel proteomic, transcriptomic and epigenomic markers (as well as other emerging -omic technologies) for CVD (i.e. aortic stenosis, cardiomyopathy, myorcardial infarction, etc). The study of physiological and genetic factors will allow for the discovery of new genomic and other -omic (including proteomic, transcriptomic and epigenomic) biomarkers associated with CVD which will lead to an improved understanding of the underlying biology of CVD and may provide future insights into the prevention and treatment of this type of disease.

DETAILED DESCRIPTION:
Inherited from parents, DNA is organized into genes and is unique to each individual. Genes contain the information that dictates how cells function and hence, can also influence the risk of developing diseases. Due to the uniqueness and variability between each individual, genes can confer different risks of developing diseases when comparing one person to another person (or a group of people). When a biological product can be measured to predict whether someone is at a higher risk for a certain disease, it is called a "biomarker". Biomarkers include, but are not limited to genetic material (such as DNA) and certain proteins found in the heart and the blood. By studying genes and proteins isolated from biological samples (blood, saliva and heart tissue), investigators of this Biobank hope to characterize known biomarkers, identify novel biomarkers and ultimately, improve the diagnosis and treatment of heart diseases.

The purpose of this research is to: (1) perform a genetic study of cardiovascular diseases, such as aortic valve diseases and (2) create a biobank (that will include blood samples, genetic material, and tissue explanted at surgery) to be used for analysis in the future.

ELIGIBILITY:
Inclusion Criteria:

* CVD diagnosis including, but not limited to: Aortic Stenosis, Coronary Heart Disease, Heart Failure, Atrial Fibrilation, Dilated Cardiomyopathy, Myocardial Infarction, and Spontaneous Coronary Artery Dissection.
* Undergoing cardiac surgery for non-aortic valve pathology

Exclusion Criteria:

* Individuals with Congenital heart disease will be excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals over 18 who meet the inclusion criteria for either the case or the control group.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
TOmAS | 5 years
  Identifying genetic differences between cases and controls.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided